CLINICAL TRIAL: NCT02213978
Title: A Clinical Cohort Study of Safety and Effectiveness of Venous Thromboembolism Prophylaxis in Critical Ill Patients
Acronym: VTEH
Status: Completed | Type: Observational
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Xiao Tang, doctor of the department of respiratory and critical care medicine of Beijing Chao Yang Hospital, Beijing Chao Yang Hospital
Other Study IDs: ICU-VTE-2014
Record Dates: First submitted 2014-08-07; First posted 2014-08-12 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Venous Thromboembolism; Hemorrhage
MeSH Terms: conditions — Venous Thromboembolism; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to analyze the effect of the prophylaxis of venous thromboembolism in the critical ill patients, and at the same time, to find out the risk of venous thromboembolism and hemorrhage events occurred under the prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* all the patients in ICUs estimated time in ICU mare than 48h

Exclusion Criteria:

* estimated time in ICU less than 48h refused to attend

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the critical ill patients in ICUs
Sampling Method: Non-Probability Sample
Enrollment: 1114 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
the incidence of venous thromboembolism under the thromboprophylaxis in critical ill patients | 2 weeks
  at the same time, to analyze the risk factor of the occurrence of venous thromboembolism despite of thromboprophylaxis

SECONDARY OUTCOMES:
the incidence of bleeding events under thromboprophylaxis in critical ill patients | 2 weeks
  at the same time, to analyze the risk factors of bleeding in critical ill patients who receive thromboprophylaxis

OTHER OUTCOMES:
the incidence of venous thromboembolism under the mechanical thromboprophylaxis in the critical ill patients who with the contraindications to anticoagulation | 2 weeks
  At the same time,to analyze the aspects below:
  1. Evaluation the tolerance to mechanical thromboprophylaxis of these patients
  2. Comparison of the effectiveness between intermittent pneumatic compression and graduated compression stockings in mechanical thromboprophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Tang, MD, Principal Investigator — Beijing Chao-Yang Hospital,China
Locations (1):
- Department of respiratory and critical care medicine,Beijing Chao-yang Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lyu WR, Tang X, Jin Y, Wang R, Li XY, Li Y, Zhang CY, Zhao W, Tong ZH, Sun B. Hemorrhages and risk factors in patients undergoing thromboprophylaxis in a respiratory critical care unit: a secondary data analysis of a cohort study. J Intensive Care. 2024 Oct 29;12(1):43. doi: 10.1186/s40560-024-00756-w. PMID 39473017
- [Derived] Tang X, Lyu WR, Jin Y, Wang R, Li XY, Li Y, Zhang CY, Zhao W, Tong ZH, Sun B. Modern thromboprophylaxis protocol based on guidelines applied in a respiratory intensive care unit: a single-center prospective cohort study. Thromb J. 2022 Dec 12;20(1):76. doi: 10.1186/s12959-022-00439-2. PMID 36510234